CLINICAL TRIAL: NCT06802549
Title: Treatment Outcomes of Partial Pulpotomy Using Two Different Calcium Silicate Materials in Cariously Exposed Mature Permanent Teeth: A Randomized Clinical Trial
Brief Title: Outcomes of Partial Pulpotomy Treatment in Cariously Exposed Teeth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Tuba Gök, PhD., Assistant Professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIRATUNI-DENTISTRY-TUBAGOK-002
Record Dates: First submitted 2025-01-20; First posted 2025-01-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Deep Dental Caries
Keywords: deep dental caries; partial pulpotomy; calcium silicate-based material

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Partial Pulpotomy with Biodentine (Active Comparator)
  Interventions: Device: Biodentine (calcium silicate-based cement) (Septodont, Saint Maur de Fossés, France)
- Partial Pulpotomy with Theracal PT (Experimental)
  Interventions: Device: Theracal PT (resin modified calcium silicate-based cement) (Bisco Inc., Schaumburg, IL, USA)

INTERVENTIONS:
Device: Biodentine (calcium silicate-based cement) (Septodont, Saint Maur de Fossés, France) — It will be placed on the exposed pulp with the help of a carrier and the exposed pulp will be covered with material
  Arms: Partial Pulpotomy with Biodentine
Device: Theracal PT (resin modified calcium silicate-based cement) (Bisco Inc., Schaumburg, IL, USA) — It will be placed on the exposed pulp with the help of its injection tip and the exposed pulp will be covered with material
  Arms: Partial Pulpotomy with Theracal PT

SUMMARY:
The aim of this clinical trial is to learn how successful Biodentine and Theracal PT dental filling materials are in treating deep tooth decay in adults. It will also provide information about post-treatment pain. The main questions it aims to answer are:

Do Biodentine and Theracal PT dental filling materials treat exposed tooth decay in participants? Do they reduce the need for root canal treatment? After the application of Biodentine and Theracal PT dental filling materials to the participants, the pain and symptoms that cause pain may not decrease. In this case, the tooth may be treated with root canal treatment. The researchers will compare the clinical success of Biodentine and Theracal PT dental filling materials with each other.

Participants will undergo a single-session partial pulpotomy treatment with the dental filling materials mentioned above. Clinical and radiographic follow-ups will then be performed at 3, 6 and 12 months, and records will be kept.

ELIGIBILITY:
Inclusion Criteria:

* • Patient age should be between 18-50 years

  * Should be able to give written informed consent
  * Should have systemic status (ASA 1)
  * Should have permanent molar or premolar (lower and upper) root development
  * Should be asymptomatic, deep (D3) or extremely deep (D4) caries
  * Should give vital response in cold test and electric pulp test
  * Should have teeth where the pulp is exposed with caries
  * Should not have pain during palpation and percussion
  * Should not have periodontal disease
  * Should have restorable teeth
  * Should have teeth without pulp necrosis, sinus tract or swelling/abscess
  * Should have bleeding time less than 10 minutes
  * Should be able to include a maximum of two teeth in a patient in the study (should be in different quadrants and there should be at least 2 weeks between treatment periods)

Exclusion Criteria:

* Teeth with incomplete root development

  * Severely affected teeth that do not respond to pulp sensitivity tests
  * Teeth with signs and symptoms of irreversible pulpitis
  * Teeth without signs of bleeding after communicating with the pulp chamber
  * Teeth with pulp chamber open to the oral environment
  * Teeth with periodontal pockets greater than 4 mm deep
  * Teeth with suspected cracks or crown fractures that may be responsible for pulp pathology
  * Teeth with uncontrolled bleeding
  * Medically at-risk patients will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
"Tooth survival". Both clinical and radiographic healing means "Tooth survival". Clinical healing; absence of clinical symptoms. Radiographic healing; absence of emerging periapical radiolucency. | From enrollment to the end of treatment at 1 year

SECONDARY OUTCOMES:
"Post operative pain". It will be evaluated with a 10-unit visual analog scale. 0: no pain, 1-3 mild pain, 4-6 moderate-severe pain, 7-9 very severe pain, 10 worst pain. | From enrollment to the follow up at 1 week, 3,6.12 months"

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Title: Data Sharing for Parial Pulpotomy Treatment in Teeth with Cariously Exposed:
  The objective of this IPD (Individual Participant Data) sharing plan is to enhance the understanding of the success of partial pulpotomy treatment in cariously exposed teeth using Biodentine and Theracal PT materials, by encouraging and supporting data analysis.
  Data Access Conditions: Access to the data is available to researchers who present a valid proposal for research purposes and sign a data use agreement. All applications will be reviewed by the study management committee.
  Data Use: Data may only be used for scientific and ethical research purposes. Data Storage: Data will be stored for a period of ten years following the completion of the study and will be securely disposed of at the end of this period.
  Data Protection: Data will be stored under strict security protocols and accessible only to authorized personnel.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Duncan HF. Present status and future directions-Vital pulp treatment and pulp preservation strategies. Int Endod J. 2022 May;55 Suppl 3(Suppl 3):497-511. doi: 10.1111/iej.13688. Epub 2022 Feb 3. PMID 35080024
- [Result] Ricucci D, Siqueira JF Jr, Li Y, Tay FR. Vital pulp therapy: histopathology and histobacteriology-based guidelines to treat teeth with deep caries and pulp exposure. J Dent. 2019 Jul;86:41-52. doi: 10.1016/j.jdent.2019.05.022. Epub 2019 May 21. PMID 31121241
- [Result] European Society of Endodontology (ESE) developed by:; Duncan HF, Galler KM, Tomson PL, Simon S, El-Karim I, Kundzina R, Krastl G, Dammaschke T, Fransson H, Markvart M, Zehnder M, Bjorndal L. European Society of Endodontology position statement: Management of deep caries and the exposed pulp. Int Endod J. 2019 Jul;52(7):923-934. doi: 10.1111/iej.13080. PMID 30664240

DOCUMENTS (2):
  • Study Protocol (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT06802549/Prot_000.pdf
  • Informed Consent Form (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT06802549/ICF_001.pdf